CLINICAL TRIAL: NCT05799989
Title: Catheter Dislocation and the Influence of Different Catheter Fixation in Pediatric Patients: Prospective Observational Trial
Brief Title: Catheter Dislocation and the Influence of Different Catheter Fixation in Pediatric Patients
Acronym: FIXATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR FIXATION 2023
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Catheter Complications
Keywords: intravenous; intraarterial; catheter; fixation; withdrawal; dislocation
MeSH Terms: conditions — Joint Dislocations | interventions — Surgical Fixation Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical fixation: Pediatric patients with intravenous and/or intraarterial catheter in situ secured with surgical fixation
  Interventions: Procedure: Surgical fixation
- Atraumatic fixation: Pediatric patients with intravenous and/or intraarterial catheter in situ secured with surgical fixation
  Interventions: Procedure: Atraumatic fixation

INTERVENTIONS:
Procedure: Surgical fixation — Pediatric patients with intravenous and/or intraarterial catheter in situ secured with surgical fixation
  Groups: Surgical fixation
Procedure: Atraumatic fixation — Pediatric patients with intravenous and/or intraarterial catheter in situ secured with atraumatic fixation
  Groups: Atraumatic fixation

SUMMARY:
Insertion of intravenous or intra-arterial catheter is one of the most common procedures in anesthesiology and intensive care medicine. After successful insertion, proper catheter fixation is required to maintain the catheter correct position with the aim to preserve catheter patency, prevent excessive movements of catheter or even iatrogenic catheter extraction/dislocation. Beside the historically preferred surgical fixation to the skin of the patient (invasive method, repeated percutaneous punction), atraumatic fixation by special dressing is currently available in clinical practice. In pediatric patients, due to limited cooperation, higher risk of dislocation exists.

DETAILED DESCRIPTION:
Pediatric patients with intravenous and/or intraarterial catheters with estimated length of insertion over 72 hours will be included into the trial.Type of catheter fixation (surgical versus atraumatic) will be evaluated. Demographic data, local and systemic complication between the group of surgical fixation and atraumatic fixation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with intravenous/intraarterial catheter secured at Departement of pediatric anesthesiology and intensive care medicine
* estimated length of catheter left in place longer than 72 hours

Exclusion Criteria:

* estimated length of catheter left in place shorter than 72 hours
* impossible patient´s evaluation after catheter insertion

Max Age: 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: pediatric patients with intravenous/intraarterial catheter secured at Departement of pediatric anesthesiology and intensive care medicine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter extraction/dislocation | In 30 days after catheter insertion
  The incidence of catheter extraction/dislocation will be evaluated between the group of surgical and atraumatic catheter fixation

SECONDARY OUTCOMES:
Incidence of local infectious complications | In 30 days after catheter insertion
  The incidence of local infectious complications will be evaluated between the group of surgical and atraumatic catheter fixation
Incidence of systemic infectious complications | In 30 days after catheter insertion
  The incidence of systemic infectious complications will be evaluated between the group of surgical and atraumatic catheter fixation
Incidence of thrombotic complications | In 30 days after catheter insertion
  The incidence of thrombotic complications will be evaluated between the group of surgical and atraumatic catheter fixation

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital - Academic Centre for Malignant Hyperthermia of Masaryk University Brno, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided